CLINICAL TRIAL: NCT01412151
Title: Creatine Safety & Tolerability in Huntington's Disease (CREST-X): A Single-Center, Open-Label, Long-Term Safety & Tolerability Extension Study of Creatine in Subjects With HD
Brief Title: Creatine Safety & Tolerability in Huntington's Disease
Acronym: CREST-X
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven M. Hersch, Professor of Neurology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005P000530
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Results first posted 2012-12-28 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Huntington's Disease (HD)
Keywords: Symptomatic; Huntington's Disease; HD
MeSH Terms: conditions — Huntington Disease | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Creatine monohydrate (Other): single arm long-term open label follow-up
  Interventions: Drug: Creatine monohydrate

INTERVENTIONS:
Drug: Creatine monohydrate — Creatine taken twice daily for a total of 30 grams daily dosage or subject's highest tolerated dose
  Other Names: creatine, crea-pure

SUMMARY:
The purpose of this study is to extend findings from the creatine dose-finding study (CREST-UP1) in Huntington's disease to evaluate the long-term safety, tolerability, and clinical impact of high dose creatine.

DETAILED DESCRIPTION:
PRÉCIS Protocol Title Creatine Safety & Tolerability in Huntington's Disease (CREST-X): A Single-Center, Open-Label, Long-Term Safety & Tolerability Extension Study of Creatine in Subjects with HD

Study Phase Phase II Clinical Trial

Funding Departmental Funds

Drug Supply Provided By The Avicena Group, Inc (Palo Alto, CA)

Number of Subjects Up to 10 subjects enrolling from the creatine dose-finding study CREST-UP1 (PHRC Protocol: 2004-P-000925)

Number of Study Centers Single site

Study Period Approximately 306 weeks on study medication Approximately 310 weeks total including follow-up

Primary Objective To evaluate the long-term safety, tolerability and clinical impact of 30 grams per day of creatine.

Secondary Objective To serve as a basis for subsequent trials designed to specifically address creatine's ability to slow or halt the progression of HD

Primary Outcome Measure Primary purpose of this study is to estimate the proportion of subjects who find the drug intolerable.

Secondary Outcome Measures 1. Changes in UHDRS subscores

2. Biological indicators that creatine might affect neuroprotection (serum creatine levels, absolute brain creatine concentrations) Significance/Relevance Several studies in rat and transgenic mouse models of HD have suggested that creatine may be neuroprotective. Most data on safety and tolerability of creatine have been performed in healthy athletes. Significant side effects were not found in studies of 14 days duration or less, while significant improvements in motor function have been shown in some studies of athletes, but not in others. There has been little data on safety and tolerability of creatine in disease conditions. In a Phase II study with HD subjects, we have found that 8g/day creatine taken over 16 weeks has been safe & well tolerated.

Study Population All subjects enrolled in CREST-UP1 who continue to meet inclusion criteria are eligible. These are men and women >18 years if age with a clinical diagnosis of HD will be considered. Sexually active women of childbearing potential may participate if they have a negative pregnancy test at screening and either use adequate birth control, are post-menopausal or are surgically sterile.

Study Design Open-label safety and tolerability study in subjects with HD enrolled at 1 site to receive creatine for approximately 306 weeks. All subjects enrolled in CREST-UP1 will be eligible to rollover into this study after the de-escalation phase; these subjects will receive 30 grams/day of creatine.

Eligibility Criteria Inclusion Criteria Subjects from CREST-UP1 eligible to continue on creatine in this extension study.

Subjects in Stage 1-3 of illness. Age of 18 years or older. Women of childbearing potential (i.e., those pre-menopausal or not surgically sterile) must confirm to the best of their knowledge that they are not pregnant or plan to get pregnant. Women of childbearing potential must have negative pregnancy test, be non-lactating and use adequate contraception methods. Adequate contraception methods include: oral birth control pills plus a barrier method (i.e. condoms, diaphragm), IUD or abstinence during the study. Abstinence will be considered an adequate contraception method on a case-to-case basis per site investigator's clinical assessment.

Subjects currently taking psychotropic medications (including antidepressants and neuroleptics) must be on stable dosages for at least 4 weeks prior to enrollment and should be maintained on constant dosage throughout the study. If clinical conditions mandate modifications of such medications, these changes will be systematically recorded and subject permitted to remain in the trial.

Subjects must be capable of providing informed consent and complying with trial procedures.

Subjects must be able to take oral medication. A person willing and able to serve as an informant and provide information about the daily dosing of study medication (if available).

Exclusion Criteria History of known sensitivity or intolerability to creatine. Subjects with underlying hematologic, hepatic or renal disease; screening white blood cell (WBC) count less than 3,800/mm3, screening creatinine greater than 2.25 or alanine aminotransferase (ALT) greater than 2 times the upper limit of normal.

Clinical evidence of unstable medical illness in the investigator's judgment. History of renal impairment (moderate to severe). Unstable psychiatric illness defined as psychosis (hallucinations or delusions), untreated major depression or suicidal ideation within 90 days of the Baseline visit.

Current or history of substance (alcohol or drug) abuse within 1 year of the Baseline visit.

Pregnant women, or women who are currently breast-feeding. Subjects who are unable to tolerate an MRI scan.

Study Procedures: Prior to taking part in the CREST-X trial, both subject and responsible informant (if available) will be provided with information about the study and will be given time to decide whether they wish to participate.

Eligible subjects from the CREST-UP1 study who wish to continue on creatine will be given the option of rolling into this study after the de-escalation phase; subjects who do not wish to continue on creatine in this study will follow Washout procedures according to the CREST-UP1 protocol.

At Baseline (Visit 1) informed consent will be obtained from each subject. All inclusion/exclusion criteria will be reviewed to determine continued eligibility for the extension study. Additional assessments will include: past/current medication, vital signs/body weight/EKG, pregnancy test (females), blood/urine samples for clinical safety/research labs.

All subjects will receive a dose of 30 grams/day; a 6-month supply of study drug will be dispensed.

Subjects will be contacted by telephone at Week 3 (Phone 1) to assess compliance with trial medication, document adverse events, and changes to concomitant medications.

During the on-study drug period, eligible subjects will return for in-person visits at Week 6 (Visit 2), Week 16 (Visit 3), Week 24 (Visit 4), Week 36 (Visit 5), Week 64 (Visit 6), Week 88 (Visit 7), Week 112 (Visit 8), Week 136 (Visit 9), as well as for Visits 10-15 (Weeks 25-170 post Visit 9), and/or withdrawal, for the following evaluations: general medical exam, vital signs/body weight/EKG, review of concomitant medication, study drug compliance, adverse events, and clinical safety/research labs. UHDRS will be completed at Week 24 (Visit 4), Week 64 (Visit 6), Week 88 (Visit 7), Week 112 (Visit 8), and Week 136 (Visit 9) and Visits 10-15. MRI will be completed at Week 24 (Visit 4), Week 64 (Visit 6), Week 88 (Visit 7), Week 112 (Visit 8), and Week 136 (Visit 9) and Visits 10-15. Subjects will receive a new supply of study drug approximately every three months as needed.

Intermittent assessments during the on-study drug period will be completed at Week 9 (Phone 2), Week 18 (Phone 3), Week 30 (Phone 4), Week 52 (Phone 5), Week 76 (Phone 6), Week 100 (Phone 7), and Week 124 (Phone 8) to primarily evaluate compliance with trial medication (during on-study period), document adverse events, and changes to concomitant medications.

Subjects who demonstrate unexpected long-term toxicity or who no longer wish to remain in the study will proceed to Washout and be followed for eight weeks off-study drug.

At Phone Washout 1 (approximately 172 weeks post-Visit 9 subjects will be contacted by telephone primarily to document any adverse events and changes in concomitant medication during the washout period.

At Visit Washout 1 (approximately 174 weeks post-Visit 9 subjects will return for the following evaluations: general medical exam, vital signs/body weight/EKG, UHDRS, review of concomitant medication, adverse events, and clinical safety/research labs, and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have completed the CREST-UP1 study.
* Individuals who are able to take oral medication.
* Individuals capable of providing informed consent and complying with trial procedures.

Exclusion Criteria:

* History of known sensitivity or intolerability to creatine.
* Clinical evidence of unstable medical illness in the investigator's judgment.

Additional eligibility criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Rosas, MD, MS, Principal Investigator — Massachusetts General Hospital; Steven M Hersch, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- [Background] Hersch SM, Gevorkian S, Marder K, Moskowitz C, Feigin A, Cox M, Como P, Zimmerman C, Lin M, Zhang L, Ulug AM, Beal MF, Matson W, Bogdanov M, Ebbel E, Zaleta A, Kaneko Y, Jenkins B, Hevelone N, Zhang H, Yu H, Schoenfeld D, Ferrante R, Rosas HD. Creatine in Huntington disease is safe, tolerable, bioavailable in brain and reduces serum 8OH2'dG. Neurology. 2006 Jan 24;66(2):250-2. doi: 10.1212/01.wnl.0000194318.74946.b6. PMID 16434666
- [Background] Kim J, Amante DJ, Moody JP, Edgerly CK, Bordiuk OL, Smith K, Matson SA, Matson WR, Scherzer CR, Rosas HD, Hersch SM, Ferrante RJ. Reduced creatine kinase as a central and peripheral biomarker in Huntington's disease. Biochim Biophys Acta. 2010 Jul-Aug;1802(7-8):673-81. doi: 10.1016/j.bbadis.2010.05.001. Epub 2010 May 9. PMID 20460152
- [Background] Rosas HD, Salat DH, Lee SY, Zaleta AK, Pappu V, Fischl B, Greve D, Hevelone N, Hersch SM. Cerebral cortex and the clinical expression of Huntington's disease: complexity and heterogeneity. Brain. 2008 Apr;131(Pt 4):1057-68. doi: 10.1093/brain/awn025. Epub 2008 Mar 12. PMID 18337273
- [Background] Dedeoglu A, Kubilus JK, Yang L, Ferrante KL, Hersch SM, Beal MF, Ferrante RJ. Creatine therapy provides neuroprotection after onset of clinical symptoms in Huntington's disease transgenic mice. J Neurochem. 2003 Jun;85(6):1359-67. doi: 10.1046/j.1471-4159.2003.01706.x. PMID 12787055
- [Background] Stack EC, Dedeoglu A, Smith KM, Cormier K, Kubilus JK, Bogdanov M, Matson WR, Yang L, Jenkins BG, Luthi-Carter R, Kowall NW, Hersch SM, Beal MF, Ferrante RJ. Neuroprotective effects of synaptic modulation in Huntington's disease R6/2 mice. J Neurosci. 2007 Nov 21;27(47):12908-15. doi: 10.1523/JNEUROSCI.4318-07.2007. PMID 18032664
- [Background] Hersch SM, Rosas HD. Neuroprotective therapy for Huntington's disease: new prospects and challenges. Expert Rev Neurother. 2001 Sep;1(1):111-8. doi: 10.1586/14737175.1.1.111. PMID 19811052
- [Background] Borovecki F, Lovrecic L, Zhou J, Jeong H, Then F, Rosas HD, Hersch SM, Hogarth P, Bouzou B, Jensen RV, Krainc D. Genome-wide expression profiling of human blood reveals biomarkers for Huntington's disease. Proc Natl Acad Sci U S A. 2005 Aug 2;102(31):11023-8. doi: 10.1073/pnas.0504921102. Epub 2005 Jul 25. PMID 16043692
- [Background] Ryu H, Rosas HD, Hersch SM, Ferrante RJ. The therapeutic role of creatine in Huntington's disease. Pharmacol Ther. 2005 Nov;108(2):193-207. doi: 10.1016/j.pharmthera.2005.04.008. Epub 2005 Aug 1. PMID 16055197
- [Background] Hersch SM, Rosas HD. Neuroprotection for Huntington's disease: ready, set, slow. Neurotherapeutics. 2008 Apr;5(2):226-36. doi: 10.1016/j.nurt.2008.01.003. PMID 18394565
- [Background] Rosas HD, Salat DH, Lee SY, Zaleta AK, Hevelone N, Hersch SM. Complexity and heterogeneity: what drives the ever-changing brain in Huntington's disease? Ann N Y Acad Sci. 2008 Dec;1147:196-205. doi: 10.1196/annals.1427.034. PMID 19076442

RESULTS

PARTICIPANT FLOW:
Groups:
- Creatine Monohydrate: Twice daily with a meal mixed in a liquid for a total daily dosage of 30 grams. Daily dosage adjustments (e.g. reductions, suspensions, rechallenges) were allowed to manage adverse events.
Period: Week 0 - 306 - Treatment Period
Arm/Group | Creatine Monohydrate
Started | 10
Completed | 5
Not Completed | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by Investigator | 3
Period: Week 306 - 310 - Washout Period
Arm/Group | Creatine Monohydrate
Started | 5
Completed | 3
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Creatine Monohydrate
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Tolerability
Description: Proportion of subjects able to complete treatment
Time Frame: 306 Weeks
Measure: Number; unit: Participants
Arm/Group | Creatine Monohydrate
Number analyzed (Participants) | 10
Participants | 5

2. Secondary Outcome: Clinical Measures Resources Not Available to Complete Secondary Analyses.
Description: Components of the UHDRS (Unified Huntington Disease Rating Scale)
  data was not collected or analyzed for this outcome measure.
Time Frame: 310 Weeks
Population: data was not collected or analyzed for this outcome measure.
Groups:
- Creatine Monohydrate: Creatine monohydrate: Creatine taken twice daily for a total of 30 grams daily dosage or subject's highest tolerated dose.
  Data not analyzed.
Arm/Group | Creatine Monohydrate
Number analyzed (Participants) | 0

3. Secondary Outcome: Biological Markers of Disease Progression
Description: Biological indicators that creatine treatment might affect the progression of HD: serum creatine levels, neuroimaging, metabolomic and gene expression analysis
Time Frame: 310 Weeks
Population: data was not collected or analyzed for this outcome measure.
Arm/Group | Creatine Monohydrate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 310 Weeks
Description: Adverse events were assessed clinically (symptoms reported by the subject or signs detected on examination/through ancillary testing - vital signs, EKG, laboratory tests etc). Stable chronic conditions (e.g. diabetes, arthritis) present prior to the start of the study that did not worsen during the trial were not considered adverse events.
Arm/Group | Creatine Monohydrate
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creatine Monohydrate (N=10)
Agitation (Psychiatric disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Depression with Suicidal Ideation (Psychiatric disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creatine Monohydrate (N=10)
Agitation (Psychiatric disorders) | 5 (9)
Fall (Injury, poisoning and procedural complications) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Infection (Infections and infestations) | 1 (5)

LIMITATIONS AND CAVEATS:
secondary analyses no completed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No